CLINICAL TRIAL: NCT06909812
Title: A Observer Blind Randomized Controlled Pilot Trial to Determine the Equivalence of a Silicone Gel With Superoxidized Water vs. a Pirfenidone Gel for the Treatment of Hypertrophic Scars and Keloids
Brief Title: Silicone vs Pirfenidone in the Treatment of Hypertrophic Scars and Keloids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Nacional para la Enseñanza y la Investigación de la Dermatología A.C. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNEIDAC_Keloids_K131672
Record Dates: First submitted 2015-07-30; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Scars; Keloids; Hypertrophic Scar
Keywords: scars; keloids; hyperthrophic; pirfenidone
MeSH Terms: conditions — Cicatrix; Keloid; Cicatrix, Hypertrophic | interventions — pirfenidone; Gels

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Tubes containg both active treatments were identical. Outcomes assessor was blinded to treatment arm.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Silicone Gel (Active Comparator): A gel containing silicone
  Interventions: Drug: silicon gel
- Topical Pirfenidone Gel (Active Comparator): A gel containing pirfenidone
  Interventions: Drug: pirfenidone 8% gel

INTERVENTIONS:
Drug: pirfenidone 8% gel — topic aplication
  Other Names: kitoscell
  Arms: Topical Pirfenidone Gel
Drug: silicon gel — topic aplication
  Other Names: Kelodacyn
  Arms: Topical Silicone Gel

SUMMARY:
Justification:

Keloid scars are a major medical and cosmetic problem, especially in darker skin types that predominate in Mexico. It is estimated that hypertrophic scars affecting from 1.5 to 4.5% of the general population. However, the exact prevalence is unknown but studies show that going from 32 to 67%. And there are studies documenting that this prevalence is higher in Hispanic and black individuals and in the pediatric population.

Keloid scars can become highly symptomatic disfiguring and which affects the quality of life of patients and their self-esteem.Problem Statement:

Is silicone gel solutions superoxidation with equal or better than the gel 8% pirfenidone to treat keloids and hypertrophic scars?

Goal:

To evaluate the efficacy of a silicone gel-oxidation with solutions compared to a gel containing 8% pirfenidone.

Hypothesis:

If the silicone gel solutions superoxidation is equal or better than gel 8% pirfenidone to treat keloids and hypertrophic scars, then the reduction in the ECV and the EVA will be similar in the first group than the second.

Design:

Comparative, observer blind, experimental and prospective study.

DETAILED DESCRIPTION:
This is a comparative, non-inferiority, experimental, prospective, longitudinal pilot study with blind evaluator, in patients with keloid or hypertrophic scars. Twenty patients per group randomly assigned to receive identical tubes of either a silicone-based gel with superoxidized water, or an 8% pirfenidone gel. Follow-up was scheduled at 2, 4, 8, 12, and 16 weeks recording the location, mechanism of the scar, time of evolution, skin phototype, accompanying symptoms, Dermatology Life Quality Index, and validated scar assessment tools (Patient and Observer Scar Assessment Scale, Vancouver Scar Scale, and the Analog Visual Scale for Keloids).

ELIGIBILITY:
Inclusion Criteria:

* keloid or hypetrophic scar

Exclusion Criteria:

* collagen diseases pregnancy previous treatment for 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
Dermatology Life Quality Index Score | 3 months
  A life quality index for dermatological conditions
Patient and Observer Scar Assessment Scale Score | 3 months
  A validated scale (POSAS and OSAS) to assess relevant clinical characteristics of scars.
Vancouver Scar Scale | 3 months
  A validated scar scale

CONTACTS AND LOCATIONS:
Overall Officials: Jose Contreras-Ruiz, Principal Investigator — Hospital General Dr Manuel Gea Gonzalez
Locations (1):
- Hospital General Manuel Gea González, Mexico City, Mexico City, Mexico